CLINICAL TRIAL: NCT05133713
Title: Ventilation and Perfusion Imaging in Acute Pulmonary Embolism Following Catheter Directed Aspiration Thrombectomy Versus Conservative Therapy Alone: A Pilot Study
Brief Title: Ventilation and Perfusion Scan in Pulmonary Embolism Following Catheter Directed Thrombectomy Versus Anticoagulation Alone
Acronym: VQPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: Inari Medical (Industry)
Responsible Party: Principal Investigator, Gregory Woodhead, Assistant Professor, University of Arizona
Other Study IDs: STUDY00000091
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Embolism; Pulmonary Hypertension; Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Embolism; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Catheter directed thrombectomy
  Interventions: Device: Catheter directed therapy; Drug: Systemic anticoagulation
- Systemic anticoagulation
  Interventions: Drug: Systemic anticoagulation

INTERVENTIONS:
Device: Catheter directed therapy — Thrombectomy
  Groups: Catheter directed thrombectomy
Drug: Systemic anticoagulation — Conservative therapy

SUMMARY:
Clinical presentation of acute pulmonary embolism (PE) is complex and varied and not uncommonly involves respiratory failure with dyspnea or hypoxia. Patients with persisting signs of respiratory failure despite anticoagulation, may benefit from catheter directed thrombectomy. Additionally, patient who receive thrombectomy are likely to have a lower residual thrombus burden measurable by ventilation-perfusion (V/Q) scan, and thereby less likely to develop chronic sequela, including chronic thromboembolic pulmonary hypertension (CTEPH) and post PE syndrome.

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) is a common disease with variable presentation and clinical outcomes. Chronic sequelae including chronic thromboembolic pulmonary hypertension (CTEPH) and post-PE syndrome are common pathologies for patient who survive the already significant inpatient mortality, and have a significant impact on both quality of life and life expectancy. To date, the ELOPE trial is the only study to prospectively compare quality of life (QoL) and dyspnea measures and six-minute walk distance (6MWD) to cardiopulmonary exercise test, revealing worse post-PE syndrome in select populations, however this study is limited to a single arm that received anticoagulation alone. New catheter directed therapies, developed in response to such poor outcomes, provide treatment options for acute PE patients when first line therapies including anticoagulation are contraindicated or have failed.

Long term studies utilizing imaging have shown a majority of patients diagnosed with PE have residual pulmonary thrombi after 6 months, which is likely to be a large contributor to the development of CTEPH. Ventilation-perfusion (V/Q) scans remain the gold standard for detection of both acute and chronic pulmonary embolism and will serve as a primary outcome measure at 6 months post initial treatment. Clinical measures including 6MWD, QoL and dyspnea questionaries will be assessed prior to discharge, and at 1 and 6 months, in order to characterize the development of chronic symptomatology.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Clinical signs and symptoms consistent with acute PE
3. Echocardiogram, CT pulmonary angiogram (CTPA) or pulmonary angiographic evidence of proximal filling defect in at least one main or lobar pulmonary artery
4. Scheduled for PE treatment with catheter directed therapy and systemic anticoagulation or anticoagulation alone per the investigator's discretion
5. Signs of respiratory failure including a. arterial blood saturation <90%, or b. partial arterial oxygen pressure <60 mmHg, or c. persistent tachypnea with respiratory rates > 20/min

Exclusion Criteria:

1. Unable to be anticoagulated with heparin or alternative therapy
2. Diagnosis with a minor PE without signs of right ventricular (RV) dysfunction
3. Known sensitivity to radiographic contrast agents that, in the Investigator's opinion, cannot be adequately pre-treated
4. Imaging evidence or other evidence that suggests, in opinion of the Investigator, the patient is not appropriate for mechanical thrombectomy intervention (e.g., inability to navigate to target location or predominately chronic clot)
5. Life expectancy <6 months, as determined by the Investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients requiring treatment for acute pulmonary embolism.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation-perfusion mismatch | 6 months
  Mismatch on ventilation-perfusion scintigraphy per Prospective Investigation of Pulmonary Embolism Diagnosis (PIOPED) criteria

SECONDARY OUTCOMES:
6-minute walk distance | 30 days
6-minute walk distance | 6 months
Hospital length of stay | Up to 30 days
Dyspnea questionnaire | up to 72 hours
Dyspnea questionnaire | 30 days
Dyspnea questionnaire | 6 months
Quality of life questionnaire | 30 days
Quality of life questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldhaber SZ, Visani L, De Rosa M. Acute pulmonary embolism: clinical outcomes in the International Cooperative Pulmonary Embolism Registry (ICOPER). Lancet. 1999 Apr 24;353(9162):1386-9. doi: 10.1016/s0140-6736(98)07534-5. PMID 10227218
- [Background] Casazza F, Becattini C, Bongarzoni A, Cuccia C, Roncon L, Favretto G, Zonzin P, Pignataro L, Agnelli G. Clinical features and short term outcomes of patients with acute pulmonary embolism. The Italian Pulmonary Embolism Registry (IPER). Thromb Res. 2012 Dec;130(6):847-52. doi: 10.1016/j.thromres.2012.08.292. Epub 2012 Aug 24. PMID 22921592
- [Background] Piazza G, Goldhaber SZ. Chronic thromboembolic pulmonary hypertension. N Engl J Med. 2011 Jan 27;364(4):351-60. doi: 10.1056/NEJMra0910203. No abstract available. PMID 21268727
- [Background] Kahn SR, Akaberi A, Granton JT, Anderson DR, Wells PS, Rodger MA, Solymoss S, Kovacs MJ, Rudski L, Shimony A, Dennie C, Rush C, Hernandez P, Aaron SD, Hirsch AM. Quality of Life, Dyspnea, and Functional Exercise Capacity Following a First Episode of Pulmonary Embolism: Results of the ELOPE Cohort Study. Am J Med. 2017 Aug;130(8):990.e9-990.e21. doi: 10.1016/j.amjmed.2017.03.033. Epub 2017 Apr 8. PMID 28400247
- [Background] Nijkeuter M, Hovens MM, Davidson BL, Huisman MV. Resolution of thromboemboli in patients with acute pulmonary embolism: a systematic review. Chest. 2006 Jan;129(1):192-7. doi: 10.1378/chest.129.1.192. PMID 16424432
- [Background] Kahn SR, Hirsch AM, Akaberi A, Hernandez P, Anderson DR, Wells PS, Rodger MA, Solymoss S, Kovacs MJ, Rudski L, Shimony A, Dennie C, Rush C, Geerts WH, Aaron SD, Granton JT. Functional and Exercise Limitations After a First Episode of Pulmonary Embolism: Results of the ELOPE Prospective Cohort Study. Chest. 2017 May;151(5):1058-1068. doi: 10.1016/j.chest.2016.11.030. Epub 2016 Dec 6. PMID 27932051